CLINICAL TRIAL: NCT06952517
Title: Efficacy and Safety of Topical Clascoterone Cream 1% in Patients With Facial Acneiform Rosacea
Brief Title: Efficacy and Safety of Topical Clascoterone (WINLEVI) Cream 1% in Patients With Facial Acneiform Rosacea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Narrows Institute for Biomedical Research (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1760535
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Papular-pustular Rosacea; Papulopustular Rosacea (PPR); Papulopustular Rosacea
Keywords: rosacea; papulopustular rosacea; acneiform rosacea; PPR
MeSH Terms: conditions — Rosacea | interventions — Clascoterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with Acneiform or Papulopustular Rosacea (Experimental): Patients with diagnosis of papulopustular or acneiform rosacea
  Interventions: Drug: Clascoterone Cream 1%

INTERVENTIONS:
Drug: Clascoterone Cream 1% — Clascoterone 1% cream
  Other Names: WINLEVI

SUMMARY:
To demonstrate the efficacy of Clascoterone cream 1% in reducing the size of sebaceous glands in study participants with acneiform rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18+.
* Diagnosis of rosacea type 2 (papulopustular).
* Available and willing to comply with study instructions and attend all study visits.
* Able and willing to provide written and verbal informed consent.
* Subject has used the same type and brand of make-up, other facial products, and hair products (e.g., shampoo, gel, hair spray, mousse, etc.) for at least one month prior to the baseline visit and agrees to continue his/her other general skin and hair care products and regimen for the entire study.

Exclusion Criteria:

* Subject has any skin pathology or condition that could interfere with the evaluation of the test products or requires the use of interfering topical or systemic therapy.
* Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
* Pregnant, lactating, or is planning to become pregnant during the study.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or has been treated with an investigational device within 30 days prior to the initiation of treatment (baseline).
* Study participant has facial hair that could interfere with the study assessments in the opinion of the investigator.
* Study participant is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
* Subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.
* Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Biopsy proven reduction in size of sebaceous glands at the end of 12 weeks of treatment compared to the baseline. | From enrollment to end of treatment at 12 weeks
  We will perform both a paired and pooled statistical analysis. We will conduct a power analysis to determine statistical significance. For the paired analysis, we will calculate the average gland size per patient at baseline and again at the end of the treatment period from all the individual's biopsy sites. We will then calculate the percent reduction of sebaceous gland size between the two average sizes. Finally, we will calculate the average percent change across all participants.
  For the pooled analysis, we will calculate the average sebaceous gland size across all study participants before and after treatment. We will use these two values to calculate the percent change. We anticipate that the paired analysis will yield more meaningful results as the pooled analysis may not show significant change due to the variations between study participants used to calculate the averages.

SECONDARY OUTCOMES:
Evaluation of safety and adverse events | From enrollment to end of treatment at 12 weeks
  We plan to calculate the incidence of adverse events. Study participants will be instructed to keep a log of all adverse events.
Pre- and post-treatment digital photography with a camera (Canfield Scientific, Parsippany, NJ) to depict clinical improvement of rosacea. | From enrollment to end of treatment at 12 weeks
  Pre- and post-treatment digital photography with a camera (Canfield Scientific, Parsippany, NJ) to depict clinical improvement of rosacea.
Physician and study participants reported assessments at the end of the treatment compared to baseline | From enrollment to end of treatment at 12 weeks
  A modified, succinct version of the Rosacea clinical scorecard as proposed by the Report of the National Rosacea Society Expert Committee on the Classification and Staging of sRosacea will be used to assess these measures. Physicians and study participants will be asked to grade the rosacea at baseline and at the end of the treatment based on the following scale:
  * Subtype 1: Erythematotelangiectatic: 1=Absent, 2=Mild, 3=Moderate, 4=Severe
  * Subtype 2: Papulopustular: 1=Absent, 2=Mild, 3=Moderate, 4=Severe
  * Subtype 3: Phymatous: 1=Absent, 2=Mild, 3=Moderate, 4=Severe
  * Global Assessment: 1=Absent, 2=Mild, 3=Moderate, 4=Severe

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD MS, Principal Investigator — SUNY Downstate Health Sciences University Department of Dermatology
Locations (1):
- New York Harbor VA Brooklyn Campus, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD may not be shared because this study is conducted at a VA hospital with a small sample size

REFERENCES:
- [Background] Liakou AI, Nyengaard JR, Bonovas S, Knolle J, Makrantonaki E, Zouboulis CC. Marked Reduction of the Number and Individual Volume of Sebaceous Glands in Psoriatic Lesions. Dermatology. 2016;232(4):415-24. doi: 10.1159/000445942. Epub 2016 Jun 2. PMID 27250651
- [Background] Wilkin J, Dahl M, Detmar M, Drake L, Liang MH, Odom R, Powell F; National Rosacea Society Expert Committee. Standard grading system for rosacea: report of the National Rosacea Society Expert Committee on the classification and staging of rosacea. J Am Acad Dermatol. 2004 Jun;50(6):907-12. doi: 10.1016/j.jaad.2004.01.048. No abstract available. PMID 15153893
- [Background] Buhl T, Sulk M, Nowak P, Buddenkotte J, McDonald I, Aubert J, Carlavan I, Deret S, Reiniche P, Rivier M, Voegel JJ, Steinhoff M. Molecular and Morphological Characterization of Inflammatory Infiltrate in Rosacea Reveals Activation of Th1/Th17 Pathways. J Invest Dermatol. 2015 Sep;135(9):2198-2208. doi: 10.1038/jid.2015.141. Epub 2015 Apr 7. PMID 25848978
- [Background] Brelsford M, Beute TC. Preventing and managing the side effects of isotretinoin. Semin Cutan Med Surg. 2008 Sep;27(3):197-206. doi: 10.1016/j.sder.2008.07.002. PMID 18786498
- [Background] Khalil NY, Darwish IA, Al-Qahtani AA. Isotretinoin. Profiles Drug Subst Excip Relat Methodol. 2020;45:119-157. doi: 10.1016/bs.podrm.2019.10.005. Epub 2019 Dec 6. PMID 32164966
- [Background] Tan J, Schofer H, Araviiskaia E, Audibert F, Kerrouche N, Berg M; RISE study group. Prevalence of rosacea in the general population of Germany and Russia - The RISE study. J Eur Acad Dermatol Venereol. 2016 Mar;30(3):428-34. doi: 10.1111/jdv.13556. PMID 26915718